CLINICAL TRIAL: NCT05173948
Title: Effectiveness of Kinesio Taping and Conventional Physical Therapy in the Management of Chronic Low Back Pain
Brief Title: The Effectiveness of Kinesio Taping in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tabuk (Other)
Responsible Party: Principal Investigator, Shahul Hameed Pakkir Mohamed, Assistant Professor, University of Tabuk
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UT-79-11-2019
Record Dates: First submitted 2021-11-23; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Chronic Low-back Pain
Keywords: Low back pain; Chronic; Kinesio taping; TENS; Exercises
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping and Conventional Physical therapy (Experimental): Kinesio taping with Transcutaneous Electrical Nerve Stimulation and Supervised Exercise therapy
  Interventions: Other: Kinesio taping; Device: Conventional physical therapy
- Conventional Physical therapy (Experimental): Transcutaneous Electrical Nerve Stimulation and Supervised Exercise therapy
  Interventions: Device: Conventional physical therapy

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping: The tape is measured from the sacrum to the 12th thoracic vertebra with forwarding flexion of the trunk. The base is affixed to the insertion in the resting position. The muscle is elongated and the base anchored with skin displacement. The tape is then affixed with 10% stretch paravertebrally over the muscle bundles up to T12. The tape is rubbed with the muscle in the elongated state.
  Arms: Kinesio taping and Conventional Physical therapy
Device: Conventional physical therapy — Transcutaneous electrical nerve stimulation device settings, such as the frequency of 80 Hz, the pulse width of 100 µs, and symmetrical biphasic waveform. Four mediums sized (2 × 2 cm) carbon-impregnated rubber cutaneous electrodes were placed bilaterally in a standard dermatomal pattern over the most painful lumbar region. The current intensity was increased up to the patient's perception of paraesthesia. The supervised exercise therapy management consisted of stretching exercises for the back, iliopsoas, gluteal and hamstring muscles, and strengthening exercises for the abdominal and back muscles. Three sets of stretching exercises, each involving a 30-sec hold and 30-sec of rest repeated three times, were performed in three sessions per week over four weeks. One set of strengthening exercises, consisting of 10 repetitions with a 5-sec hold, was performed in three sessions per week over four weeks.

SUMMARY:
The objective of this study is to determine the effectiveness of Kinesio taping (KT) with Conventional Physical therapy (CPT) - Transcutaneous Electrical Nerve Stimulation (TENS) and Supervised Exercise therapy and CPT in the management of CLBP.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is one of the most common causes of chronic disability which leads to major social and economic consequences. The role and effectiveness of the Kinesio taping (KT) and Conventional Physical therapy (CPT) are evident from the existing literature but no comparison was found on the combination of other physical therapy techniques such as supervised exercise therapy and Transcutaneous Electrical Nerve Stimulation (TENS) with CLBP in the Kingdom of Saudi Arabia

ELIGIBILITY:
Inclusion Criteria:

* Pain caused by mechanical/nonspecific low back pain.
* Degeneration of the spine and intervertebral disc.
* The visual analog scale of pain 4 and above
* Low back pain for at least three months

Exclusion Criteria:

* Physical therapy treatment is taken in the past 6 months period
* Previous spinal surgery with fixation
* Structural anomalies
* Spinal cord compression
* Severe osteoporosis
* Acute infections
* Severe cardiovascular or metabolic diseases
* Pregnant women

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | Six weeks
  Pain, for the Average pain intensity over the last week was measured on a numerical pain rating scale, where 0 represented no pain and 10 represented the worst pain possible
Modified Oswestry low back pain disability questionnaire | Six weeks
  Disability were measured using the Modified Oswestry Disability Index (MODI) which is a self-rating questionnaire used to evaluate functional physical disability
Lumbar range of motion-Modified Schober test | Six weeks
  Lumbar flexion range of motion were measured by using modified Schober method

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tabuk, Tabuk, North West, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pakkir Mohamed SH, Al Amer HS, Nambi G. The effectiveness of Kinesio taping and conventional physical therapy in the management of chronic low back pain: a randomized clinical trial. Clin Rheumatol. 2023 Jan;42(1):233-244. doi: 10.1007/s10067-022-06352-3. Epub 2022 Sep 1. PMID 36045306